CLINICAL TRIAL: NCT03151031
Title: Effect on Dynamic Postural Stability After Application of Cryotherapy to the Knee Joint: A Pilot Randomized Controlled Trial
Brief Title: Effect on Dynamic Postural Stability After Application of Cryotherapy to the Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Assistant Professor, Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMIPR/SPCA/17/14
Record Dates: First submitted 2017-05-07; First posted 2017-05-12 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cryotherapy Effect; Balance; Disorder, Fluid
Keywords: balance; college students; star excursion balance test
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be informed about the reason for performing the star excursion balance test before and after the application of cryotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, the participants will be asked to perform star excursion balance test (SEBT) under two conditions, before and after the application of cryotherapy
  Interventions: Procedure: Cryotherapy
- Control Group (No Intervention): In the control group, the participants will be asked asked to perform star excursion balance test (SEBT) under two conditions, before and after 10 minutes rest

INTERVENTIONS:
Procedure: Cryotherapy — The cooling procedure for the knee joint will be initiated by using a cryopack or cold-pack. On completion of the initial SEBT, the participant will lie supine and the investigator will apply the cryotherapy for 10 minutes. After the 10 minute period of cryotherapy, the cryopack will be removed, and the participants will perform SEBT for the second time.
  Arms: Experimental Group

SUMMARY:
The purpose of this study will determine the effect of cryotherapy applied to the knee joint on static and dynamic standing balance. It is hypothesized that there will be no change in dynamic postural stability after cryotherapy application.Twenty four individuals (age 18 to 30) participated in the study. They will be randomly divided into two groups, experimental and control group. Each participant, in the experimental group will be asked to perform star excursion balance test (SEBT) under two conditions, before and after the application of cryotherapy. The participants will receive ice pack wrapping of the knee for 10 minutes. The control group performed SEBT at room temperature in an interval of 10 minutes. The two group will be analysed and compared

DETAILED DESCRIPTION:
The cooling procedure for the knee joint was initiated by using a cryopack or cold-pack. On completion of the initial SEBT, the participant lied supine and the investigator applied the cryotherapy for 10 minutes. After the 10 minute period of cryotherapy, the cryopack was removed, and the participants performed SEBT for the second time.

ELIGIBILITY:
Inclusion Criteria:

* Normal adult person.
* Aged between 18 to 30 year
* Both male and female were included in the study

Exclusion Criteria:

* Adult having any visual impairment
* Adult having any vestibular impairment
* Adult suffering from any neurological disorders
* Adult suffering from other medical conditions, like- Vascular diseases
* Adult having any disorders or conditions like- Genu valgum, Genu varum, history of knee joint or lower limb injury, or lower limb fracture

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Star Excursion Balance test at 10 minutes | Upto 10 minutes
  Distance reach in 8 directions will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Asir J Samuel, MPT, Study Director — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation
Locations (1):
- Asir John Samuel, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Through ms excel file in data repository of university
Supporting Information: Study Protocol, SAP
Time Frame: 1
Access Criteria: https://www.termedia.pl/Effect-on-dynamic-postural-stability-after-application-of-cold-therapy-to-the-knee-joint-A-pilot-randomized-controlled-trial,128,43981,0,1.html
URL: https://www.termedia.pl/Effect-on-dynamic-postural-stability-after-application-of-cold-therapy-to-the-knee-joint-A-pilot-randomized-controlled-trial,128,43981,0,1.html

REFERENCES:
- See also: Published Research — http://www.termedia.pl/Effect-on-dynamic-postural-stability-after-application-of-cold-therapy-to-the-knee-joint-A-pilot-randomized-controlled-trial,128,43981,0,1.html